CLINICAL TRIAL: NCT00904878
Title: A Multicenter National Prospective Study of Pregnancy and Neonatal Outcomes in Women With Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CCFA Pregnancy Registry; CCFA pregnancy Registry (Other: Crohn's and Colitis Foundation of America)
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Disease
Keywords: pregnant IBD patients
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A Multicenter National Prospective Study of Pregnancy and Neonatal Outcomes in Women with Inflammatory Bowel Disease study is being conducted at the University of California San Francisco and 30 other sites around the United States who are part of the CCFA Clinical Alliance. The aim of this study is to determine the effect of medication use and disease activity on the outcome of pregnancy among women with IBD up to 18 years from birth.

DETAILED DESCRIPTION:
All pregnant women with IBD diagnosis who are taking biologics medicines and immunosuppressants will be entered in the study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with confirmed IBD diagnoses who are pregnant and taking immunosuppressants and/or biologic therapy

Exclusion Criteria:

* Pregnant female patients younger than 18 years of age
* Confirmed multiple gestation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients with confirmed IBD diagnoses who are pregnant
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2007-08; Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Determine whether children born to women with IBD have higher rates of developmental delay compared to their age matched non-IBD peers, as measured by the Ages and Stages Questionnaire (ASQ-3) at ages 12, 24, 36, and 48 months | December 2014

SECONDARY OUTCOMES:
Determine whether the rate of any adverse pregnancy outcomes in a prospective national sample of women from the United States with IBD differ with respect to exposure to azathioprine/6MP or anti-TNF therapy | December 2014

OTHER OUTCOMES:
Determine whether breastfeeding impacts developmental delay, growth and infectious complications in children born to women with IBD | December 2014

CONTACTS AND LOCATIONS:
Overall Officials: Uma Mahadevan, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Please Contact Jessica Lim For Further Information Regarding Other Sites' Locations, San Francisco, California
  - University of California San Francisco, San Francisco, California

REFERENCES:
- [Derived] Mahadevan U, Long MD, Kane SV, Roy A, Dubinsky MC, Sands BE, Cohen RD, Chambers CD, Sandborn WJ; Crohn's Colitis Foundation Clinical Research Alliance. Pregnancy and Neonatal Outcomes After Fetal Exposure to Biologics and Thiopurines Among Women With Inflammatory Bowel Disease. Gastroenterology. 2021 Mar;160(4):1131-1139. doi: 10.1053/j.gastro.2020.11.038. Epub 2020 Nov 21. PMID 33227283
- [Derived] Matro R, Martin CF, Wolf D, Shah SA, Mahadevan U. Exposure Concentrations of Infants Breastfed by Women Receiving Biologic Therapies for Inflammatory Bowel Diseases and Effects of Breastfeeding on Infections and Development. Gastroenterology. 2018 Sep;155(3):696-704. doi: 10.1053/j.gastro.2018.05.040. Epub 2018 May 30. PMID 29857090